CLINICAL TRIAL: NCT04883528
Title: Protecting With ARNI Against Cardiac Consequences of Coronavirus Disease 2019
Acronym: PARACOR-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00108314
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Covid19
Keywords: sacubitril/valsartan
MeSH Terms: conditions — COVID-19 | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacubitril/valsartan (Experimental): Initial dose for patients randomized to sacubitril/valsartan (LCZ696) will be determined by the blood pressure at the time of randomization. Study treatment will be titrated to the next highest dose (dose level 2 or 3) based on blood pressure at the time of visit 2/titration visit. Dose adjustments are only allowed if indicated per protocol defined criteria and per investigator judgement of safety and tolerability.
  Sacubitril/valsartan (LCZ696) tablet with minimum dose 24/26 mg, maximum dose 97/103 mg twice daily administered orally.
  Other Name: LCZ696
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet [Entresto]
- Placebo (Placebo Comparator): Initial dose for patients randomized to sacubitril/valsartan matching placebo will be determined by the blood pressure at the time of randomization. Study treatment will be titrated to the next highest dose (dose level 2 or 3) based on blood pressure at the time of visit 2/titration visit. Dose adjustments are only allowed if indicated per protocol defined criteria and per investigator judgement of safety and tolerability.
  Sacubitril/valsartan matching placebo with minimum dose matching the 24/26 mg dose, maximum dose matching the 97/103 mg dose, administered twice daily orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet [Entresto] — sacubitril/valsartan (LCZ696) tablet with minimum dose 24/26 mg, maximum dose 97/103 mg twice daily administered orally.
  Other Names: LCZ696
  Arms: Sacubitril/valsartan
Drug: Placebo — sacubitril/valsartan matching placebo tablet with minimum dose 24/26 mg, maximum dose 97/103 mg twice daily administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of sacubitril/valsartan versus placebo on markers of cardiac injury, structure, and function among patients who recovered from acute COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a history of laboratory proven-diagnosis of COVID-19 who is 4-16 weeks from their last positive COVID-19 test
2. Systolic blood pressure ≥100 mmHg at screening
3. ≥18 years of age
4. Successful collection of baseline serum biomarkers
5. Successful completion of baseline EQ-5D questionnaire
6. Successful completion of baseline CMR study (CMR sub-study only)
7. High-sensitivity troponin T at or above the level of detection on screening labs
8. Presence of ≥1 of the following:

   1. Age ≥60
   2. History of atherosclerotic cardiovascular disease (ASCVD), including myocardial infarction, coronary artery disease, ischemic stroke/transient ischemic attack, or peripheral artery disease
   3. Diabetes mellitus (Type 1 or Type 2)
   4. Body mass index ≥35 kg/m2
   5. eGFR 30-60 ml/min/1.73m2
   6. History of atrial fibrillation/flutter

Exclusion Criteria:

1. Fever within the past 96 hours of >100.3 degrees Fahrenheit
2. Actively receiving therapy with an angiotensin-converting enzyme inhibitor (ACEI), angiotensin II receptor blocker (ARB), aliskiren, or sacubitril/valsartan
3. Last known left ventricular ejection fraction of ≤40%
4. eGFR <30 ml/min/1.73m2 on screening labs, including patients on dialysis therapy
5. Serum potassium >5.0 mEq/L on screening labs
6. Prior intolerance, allergy or angioedema to ACEI, ARB, or sacubitril/valsartan
7. Pregnant or breast-feeding
8. In women of childbearing age, unwillingness to use birth control for the duration of the study
9. History of heart transplant or durable left ventricular assist device
10. Currently implanted permanent pacemaker, defibrillator, or other device that would preclude CMR testing (CMR sub-study only)
11. Currently participating in another trial of an investigational medication or device for COVID-19.
12. Any other condition that in the judgment of the investigator would jeopardize the patient's compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Greene, MD, Principal Investigator — Duke University; G. Michael Felker, MD, MHS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greene SJ, Chambers R, Lerman JB, Harrington J, deFilippi CR, Wendell DC, Kim HW, Green CL, Butler J, Felker GM. Sacubitril/valsartan and cardiovascular biomarkers among patients with recent COVID-19 infection: The PARACOR-19 randomized clinical trial. Eur J Heart Fail. 2024 Jun;26(6):1393-1398. doi: 10.1002/ejhf.3199. Epub 2024 May 11. PMID 38733160

RESULTS

PARTICIPANT FLOW:
Groups:
- Sacubitril/Valsartan: Initial dose for patients randomized to sacubitril/valsartan (LCZ696) will be determined by the blood pressure at the time of randomization. Study treatment will be titrated to the next highest dose (dose level 2 or 3) based on blood pressure at the time of visit 2/titration visit. Dose adjustments are only allowed if indicated per protocol defined criteria and per investigator judgement of safety and tolerability.
  Sacubitril/valsartan (LCZ696) tablet with minimum dose 24/26 mg, maximum dose 97/103 mg twice daily administered orally.
  Other Name: LCZ696
  Sacubitril / Valsartan Oral Tablet [Entresto]: sacubitril/valsartan (LCZ696) tablet with minimum dose 24/26 mg, maximum dose 97/103 mg twice daily administered orally.
- Placebo: Initial dose for patients randomized to sacubitril/valsartan matching placebo will be determined by the blood pressure at the time of randomization. Study treatment will be titrated to the next highest dose (dose level 2 or 3) based on blood pressure at the time of visit 2/titration visit. Dose adjustments are only allowed if indicated per protocol defined criteria and per investigator judgement of safety and tolerability.
  Sacubitril/valsartan matching placebo with minimum dose matching the 24/26 mg dose, maximum dose matching the 97/103 mg dose, administered twice daily orally.
  Placebo: sacubitril/valsartan matching placebo tablet with minimum dose 24/26 mg, maximum dose 97/103 mg twice daily administered orally.
Period: Overall Study
Arm/Group | Sacubitril/Valsartan | Placebo
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sacubitril/Valsartan | Placebo | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Median (Full Range); unit: years] | 65 [61 to 70] | 69 [65 to 71] | 67 [61 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 17 | 21 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in High-sensitivity Troponin T
Description: An elevated level of troponin T on the high-sensitivity cardiac troponin test indicates heart muscle damage or a heart attack.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
ng/mL | 1.12 [0.99 to 1.26] | 1.01 [0.87 to 1.17]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.29, Mixed Models Analysis

2. Primary Outcome: Change From Baseline in Soluble ST2
Description: ST2 is a decoy receptor that inhibits beneficial cardioprotective effects of IL-33; such inhibition results in cardiac hypertrophy, myocardial fibrosis, and ventricular dysfunction. Measurement of soluble ST2 has utility for assessing heart failure severity and prognosis.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
ng/mL | 0.95 [0.81 to 1.10] | 0.96 [0.80 to 1.15]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.88, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline in C-reactive Peptide (CRP)
Description: CRP is a pentameric protein synthesized by the liver; its level rises in response to inflammation.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
mg/dL | 0.94 [0.68 to 1.29] | 0.87 [0.55 to 1.36]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.76, Mixed Models Analysis

4. Secondary Outcome: Change From Baseline in P1NP (Procollagen Type I N-propeptide)
Description: Serum P1NP is designated as the reference marker of bone formation in osteoporosis. Elevated markers are associated with increased bone turnover, which increases the deterioration of bone quality and the risk of fragility fracture.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/L
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
mcg/L | 0.98 [0.91 to 1.05] | 0.99 [0.91 to 1.06]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.85, Mixed Models Analysis

5. Secondary Outcome: Change From Baseline in Galectin-3
Description: Galectin-3 may be used as a diagnostic or prognostic biomarker for certain types of heart disease, kidney disease and cancer.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
ng/mL | 0.89 [0.77 to 1.02] | 0.91 [0.77 to 1.09]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.80, Mixed Models Analysis

6. Secondary Outcome: Change From Baseline in NT-proBNP (N-terminal Pro B-type Natriuretic Peptide)
Description: Higher levels of NT-proBNP indicate increased heart failure.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
pg/mL | 0.60 [0.42 to 0.85] | 1.11 [0.85 to 1.45]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.01, Mixed Models Analysis

7. Secondary Outcome: Change From Baseline in GDF-15 (Growth/Differentiation Factor-15)
Description: Highly elevated GDF-15 levels are mostly linked to pathological conditions including inflammation, myocardial ischemia, and notably cancer.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
pg/mL | 1.14 [0.98 to 1.33] | 1.00 [0.85 to 1.17]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.23, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline in IL-6 (Interleukin-6)
Description: IL-6 can be elevated with inflammation, infection, autoimmune disorders, cardiovascular diseases, and some cancers.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
pg/mL | 1.10 [0.52 to 2.36] | 1.07 [0.59 to 1.93]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.95, Mixed Models Analysis

9. Secondary Outcome: Change From Baseline in CITP (C-terminal Telopeptide of Collagen Type I)
Description: Elevated levels of CITP indicate increased bone turnover.
Time Frame: Baseline, Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
ng/mL | 0.77 [0.50 to 1.18] | 1.55 [0.98 to 2.46]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.03, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: LVEF is the amount of blood pumped out of the heart's left ventricle each time it contracts, represented as a percentage of the blood in the left ventricle that gets pumped out to the body. Normal = LVEF 50% to 70% (midpoint 60%) Mild dysfunction = LVEF 40% to 49% (midpoint 45%) Moderate dysfunction = LVEF 30% to 39% (midpoint 35%) Severe dysfunction = LVEF less than 30%.
Time Frame: Baseline, Week 12
Population: Participants who consented to this optional substudy.
Measure: Mean (95% Confidence Interval); unit: percentage of blood
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 6 | 12
percentage of blood | 0.5 [-4.7 to 5.7] | 0.5 [-1.8 to 2.8]

11. Secondary Outcome: Change From Baseline in Focal Fibrosis by Delayed-enhancement on Cardiac MRI
Time Frame: Baseline, Week 12
Population: Data not collected.
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Focal Fibrosis by Percentage of Left Ventricular Myocardial Mass on Cardiac MRI
Time Frame: Baseline, Week 12
Population: Data not collected.
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in EuroQol-5 Dimensions (EQ-5D) Utility Score
Description: The EQ-5D utility score is a value that represents a person's health state based on a set of weights that reflect their preferences. The score is anchored at 0, which represents a state as bad as death, and 1, which represents full health. Negative values can be assigned to health states that are considered worse than death.
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
score on a scale | 0.01 [-0.04 to 0.06] | 0.03 [0.00 to 0.05]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.64, Mixed Models Analysis; Least squares mean difference = -0.01, 95% CI 2-sided [-0.07 to 0.04]

14. Secondary Outcome: Change From Baseline in EuroQOL-5 Dimensions (EQ-5D) Visual Analog Scale (VAS)
Description: The EQ-5D VAS is a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sacubitril/Valsartan | Placebo
Number analyzed (Participants) | 20 | 22
score on a scale | -5.60 [-11.60 to 0.40] | 1.95 [-1.73 to 5.64]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Placebo; Test type: Superiority; p = 0.04, Mixed Models Analysis; Least squares mean difference = -7.55, 95% CI 2-sided [-14.59 to 0.52]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Sacubitril/Valsartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT04883528/Prot_SAP_000.pdf